CLINICAL TRIAL: NCT02820389
Title: Observational Study to Compare the Utilisation of CT Colonography With Optical Colonoscopy as the First Diagnostic Imaging Tool in Patients With Suspected Colorectal Cancer
Brief Title: CT Colonography as the Initial Diagnostic Imaging Tool for Patients With Suspected Colorectal Cancer
Acronym: CTCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: Colon CT study
Record Dates: First submitted 2016-06-03; First posted 2016-07-01 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Optical colonoscopy: Patients with suspected colorectal cancer will undergo optical colonoscopy as the initial imaging modality.
  Interventions: Procedure: Optical colonoscopy
- CT Colonography: Patients with suspected colorectal cancer will undergo Computed Tomography Colonography (CTC) as the initial imaging modality. Subsequent imaging might be required based on the findings from the CTC scan.
  Interventions: Procedure: CTC

INTERVENTIONS:
Procedure: Optical colonoscopy — Patients with suspected colorectal cancer in this group will undergo Optical Colonoscopy as the initial imaging modality.
  Groups: Optical colonoscopy
Procedure: CTC — Patients with suspected colorectal cancer in this group will undergo Computed Tomography Colonography (CTC) as the initial imaging modality. Subsequent imaging might be required based on the findings from the CTC scan, i.e. patients with medium to large polyps or colorectal cancer will undergo Optical Colonoscopy as the second imaging test.
  Groups: CT Colonography

SUMMARY:
This study aims to evaluate whether the use of Computed Tomography Colonography (CTC) for patients with low to intermediate risk of suspected colorectal cancer decreases overall NHS costs and waiting times whilst increasing patient satisfaction compared to clinical practice with utilisation of Optical Colonoscopy.

DETAILED DESCRIPTION:
Given the recent change in the NICE guidance for the cancer pathway referral for patients with suspected colorectal cancer (See NG12), there will be an increase in demand for optical colonoscopy. Optical colonoscopy is technically difficult, resource intensive and associated with complications; therefore the increased use of CT Colonography (CTC) should be considered as an alternative. The diagnostic efficacy of CTC, in comparison to optical colonoscopy, is well established and has been shown to be accurate for identifying malignancies and medium to large polyps (≥6mm) with a greater level of patient acceptability.

The use of CTC as the first diagnostic imaging tool would identify those patients who would benefit from further investigation (colonoscopy or flexible sigmoidoscopy) to occur on the same day, as well as ruling out those who do not require further testing. This would then ensure that colonoscopy capacity can be prioritised appropriately to support the increase in demand due to the NICE guidance changes.

ELIGIBILITY:
Inclusion Criteria:

* Every adult patient over 40 years old, presenting with constipation or alternating change in bowel habits, with a differential diagnosis of suspected colorectal cancer.

Exclusion Criteria:

* Patients presenting with anaemia;
* Patients presenting with diarrhoea only for more than 6 weeks;
* Patients presenting with rectal bleeding;
* Patients who have undergone a previous whole-colon examination in the past 6 months;
* Patients who have been referred for a whole-colon examination to follow up already diagnosed colorectal cancer;
* Patients lacking capacity to give consent or participate in the study;
* Patients already taking part in any clinical trial of an investigational medicinal product (CTIMP);
* Prisoners
* Patients who are not fluent in English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bowel symptoms consistent with suspected colorectal cancer undergoing CTC or Optical Colonoscopy as the initial imaging test.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
3-month cost analysis per patient undergoing either Optical Colonoscopy or CTC as the initial imaging modality (measured in £ per patient) | 3 months following the initial imaging modality (either CTC or Optical Colonoscopy)
  The primary outcome of this study is to investigate whether the investigation of patients with suspected colorectal cancer using CTC as the first diagnostic imaging tool is cost-saving at 3 months compared to optical colonoscopy.

SECONDARY OUTCOMES:
6-month cost analysis per patient undergoing either Optical Colonoscopy or CTC as the initial imaging modality (measured in £ per patient) | 6 months following the initial imaging modality (either CTC or Optical Colonoscopy)
  This secondary outcome aims to investigate whether the investigation of patients with suspected colorectal cancer using CTC as the first diagnostic imaging tool is cost-saving at 6 months compared to optical colonoscopy.
3-month cost-effectiveness analysis per patient undergoing either CTC or Optical Colonoscopy as the initial imaging modality (measured in £ per QALY) | 3 months following the initial imaging modality (either CTC or Optical Colonoscopy)
  This secondary objective is aimed at evaluating whether the use of CTC as the initial imaging modality for patients with suspected colorectal cancer is cost-effective at 3 months compared to the use of Optical Colonoscopy.
6-month cost-effectiveness analysis per patient undergoing either CTC or Optical | 6 months following the initial imaging modality (either CTC or Optical Colonoscopy)
  This secondary objective is aimed at evaluating whether the use of CTC as the initial imaging modality for patients with suspected colorectal cancer is cost-effective at 6 months compared to the use of Optical Colonoscopy.
Frequency of incidental findings using CTC as the initial diagnostic imaging tool (measured as a %, number of patients with incidental findings in CTC / number of CTC scans) | Day 0 (following the initial CTC scan)
  CTC has the potential to investigate other intra-abdominal organs that are not seen with optical colonoscopy. Hence, CTC scans might lead to extracolonic findings. This outcome aims to evaluate the percentage of CTC scans that lead to clinically significant findings.
Likelihood ratio of CTC as the initial diagnostic imaging tool against the optical colonoscopy in patients with initial positive CTC findings for medium to large polyps and colorectal cancer (estimated using the p-value) | 3 months
  The likelihood ratio of CTC against colonoscopy in patients with initial positive CTC findings will be assessed using Colonoscopy as the gold standard.
Time taken (measured in days) to reach a definitive diagnosis and first major treatment decision based on the the initial CTC scan in comparison to Optical Colonoscopy as the initial imaging modality. | 3 months
  This objective will measure the time elapsed from the referral to either Colonoscopy or CTC and the time: 1) the test is actually performed; 2) a definitive diagnosis is reached (Optical Colonoscopy will be considered the gold standard for patients presenting positive findings in the initial CTC); and 3) the treatment decision is reached.
Do not Attend (DNA) or On the Day Cancellation rate associated with the pathway using Colonoscopy or CTC as the initial imaging test (measured as a percentage) | Day 0 (on the day of the CTC or Optical Colonoscopy scan)
  This objective aims to estimate the Do not Attend (DNA) or On the Day Cancellation (ODC) rate associated with the pathway using Colonoscopy or CTC as the initial imaging test. Given that the bowel preparation associated with CTC is easily tolerated, it is anticipated that the increase in CTC utilisation will lead to a decrease in DNA and ODC rates.
Patient satisfaction associated with both clinical pathways (i.e. using CTC or Optical Colonoscopy as the initial imaging scan) | 3 months
  To evaluate and compare the levels of patient satisfaction associated with the two pathways: i) with CTC as the initial imaging scan; and ii) with Optical Colonoscopy as the initial imaging scan. Two patient satisfaction questionnaires (on the day and 3 months following the CTC/Optical Colonoscopy test) will be used to quantify patient satisfaction.
Patient's self perceived quality of life - measured using EQ-5D-5L questionnaire | 3 months
  This objective aims to evaluate the patient's self-perceived quality of life associated with both pathways using a standard questionnaire (EQ-5D-5L).
Cost per correctly diagnosed medium to large polyps (≥6mm) and colorectal cancer using CTC as the initial investigation (measured in £ per patient) | 3 months
  The second outcome is to evaluate the cost per correctly diagnosed medium to large polyps (≥6mm) and colorectal cancer using CTC as the initial investigation.
  For patients with positive findings on CTC (either medium to large polyps and/or CRC), optical colonoscopy will be used as the comparator to assess whether the initial diagnosis with CTC was correct.

CONTACTS AND LOCATIONS:
Overall Officials: Nyree Griffin, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No